CLINICAL TRIAL: NCT04126369
Title: Impact of Mindfulness Intervention on Quality of Life in Patients With Drug-resistant Epilepsy.
Acronym: EPIMEDIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC18.209
Record Dates: First submitted 2019-08-02; First posted 2019-10-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Drug Resistant Epilepsy
Keywords: Drug Resistant Epilepsy; mindfulness; self management
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness intervention (Experimental): 12 mindfulness sessions for 3 months (1 session per week)
  Interventions: Other: mindfulness intervention
- Psycho educative programme (Active Comparator): 12 psycho educative sessions for 3 months (1 session per week)
  Interventions: Other: psycho educative programme

INTERVENTIONS:
Other: mindfulness intervention — The mindfulness program is conducted in a group session of up to 10 people. Each session lasts 2 hours. A total of 12 sessions will be conducted by a practitioner who is specifically trained in this type of programme.
  Arms: mindfulness intervention
Other: psycho educative programme — The psycho-educational control intervention will follow the same format and structure as the mindfulness meditation intervention in terms of group format, session duration and frequency. This is a therapeutic education programme developed for several years in the neurology department of the university hospital of Lyon and Grenoble. The program follows the repository recommended by the french league against epilepsy.
  Arms: Psycho educative programme

SUMMARY:
This study evaluates a mindfulness intervention in patients with drug resistant epilepsy.

Half of participants will follow a mindfulness programme, while the other half will follow a self management programme.

DETAILED DESCRIPTION:
Drug-resistant epilepsy is associated with an alteration of the quality of life mainly related to psychiatric comorbidities (anxiety and depression). The management of these comorbidities is therefore essential in patients with drug resistant epilepsy, Ideally through non-drug management to minimize the side effects of molecules.

The goal of mindfulness interventions in pathology is to learn to better live with a chronic disease by reducing the stress resulting from the disease, by increasing benevolence towards oneself, the acceptance of the disease and reducing the ruminations linked with the pathology.

Mindfulness therefore seems to be a good way for these patients to improve the management of their emotions and thus improve their quality of life what the investigators propose to evaluate in this study.

The study consists of two phases

1. First phase: comparative randomized study (primary endpoint):

   1. After inclusion, a 2 months baseline follow-up is carry to collect the judgement criteria without intervention.
   2. At the end of this period, patients will be randomly assigned to the mindfulness intervention group or the control group with the psycho educative programme. Both programmes will takes 3 months.
   3. Then a 6-months post-intervention follow-up period for both groups

   Patients will have assessment visits every 3 months. They will also complete a daily notebook including the number of seizures they have done and a scale of their "interior weather".
2. Second phase (optional):

At the end of the first phase, patients in the control group will be able to benefit from the mindfulness programme and will be followed at the end of the programme for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Drug resistant epilepsy according to the criteria of the International League Against Epilepsy (ILAE)
* Stable therapy for at least 3 months
* No planned surgery
* Patient affiliated to social security insurance or beneficiary of social security insurance.
* Signed consent

Exclusion Criteria:

* Patient who has previously had or regularly practicing mindfulness
* Patient with psychogenic non-epileptic seizures
* Pregnant woman, breastfeeding mother, person deprived of liberty by judicial or administrative decision, person subject to legal protection
* Patient with relationship disorders related to psychosis
* Patients who are unable or unwilling to work as a group or person unable to understand the topics discussed during session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Evolution of Quality Of Life In Epilepsy-Problems questionnaire (QOLIE31-P) score. | 9 months
  The QOLIE31-P questionnaire has been developed specifically to measure the quality of life of patients with epilepsy. The score ranges from 0 to 100 points. Higher scores reflect better quality of life; lower ones, worse quality of life.
  The score of QOLIE31-P will be assess prior to intervention and then at month 3, month 6 and month 9 after the beginning of the intervention.
  Ref : Cramer JA. Van Hammee G. N132 Study Group. Maintenance of improvement in health-related quality of life during long-term treatment with levetiracetam. Epilepsy & Behavior 2003; 4:118-123.

SECONDARY OUTCOMES:
Evolution of seizures frequency | 9 months
  The number of seizures will be plot by the patient on a daily notebook throughout the study period.
Evolution of psychiatric morbidity | 9 months
  The evolution of psychiatric morbidity will be assess with the Neurological Disorders Depression Inventory for Epilepsy (NNDI-E) questionnaire The NNDIE questionnaires will be assess prior to intervention month 0 and then at month 3, month 6 and month 9 after the beginning of the intervention.
  Ref: Gilliam et al., The Lancet Neurology, 2006 Micoulaud-Franchi et al., Epilepsy and Behavior, 2015
Evolution of anxiety level | 9 months
  The evolution of anxiety level will be assess with the State Trait Anxiety Inventory (STAI) questionnaire.
  The STAI questionnaire will be assess prior to intervention month 0 and then at month 3, month 6 and month 9 after the beginning of the intervention.
  Ref : Spielberger CD, 1983. Traduction française Schweitzer MB et Paulhan I, 1990. D'après Guelfi JD (58).
Evolution of stress management | 9 months
  The evolution of stress management will be assess with the Emotion Regulation abilities Questionnaire (ERQ).
  The ERQ questionnaire will be assess prior to intervention month 0 and then at month 3, month 6 and month 9 after the beginning of the intervention.
Evolution of stress level | 9 months
  The evolution of stress will be assess with the level of cortisol salivary. The salivary cortisol level will be assess prior to intervention month 0 and then at month 3, month 6 and month 9 after the beginning of the intervention.
Evolution of self acceptance and interoception | 9 months
  The evolution of self acceptance and interoception will be assess with the Self-Compassion Scale - Short Form (SCS-SF) questionnaire.
  The SCS-SF questionnaires will be assess prior to intervention month 0 and then at month 3, month 6 and month 9 after the beginning of the intervention.
  Ref: Raes, F., Pommier, E., Neff, K. D., & Van Gucht, D. (2011). Construction and factorial validation of a short form of the Self-Compassion Scale. Clinical Psychology & Psychotherapy. 18, 250-255.
Evolution of self acceptance and interoception | 9 months
  The evolution of self acceptance and interoception will be assess with the Multidimensional Assessment of Interoceptive Awareness (MAIA) questionnaire.
  The MAIA questionnaires will be assess prior to intervention month 0 and then at month 3, month 6 and month 9 after the beginning of the intervention.
  Ref: Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A (2012) The Multidimensional Assessment of Interoceptive Awareness (MAIA). PLoS ONE 7(11)
Evolution of self acceptance and interoception | 9 months
  The evolution of self acceptance and interoception will be assess with the Five Facet Mindfulness Questionnaire (FFMQ) The FFMQ questionnaires will be assess prior to intervention month 0 and then at month 3, month 6 and month 9 after the beginning of the intervention.
  Ref: Baer, R.A., Carmody, J., & Hunsinger, M (2012) FFMQ-SF. Journal of Clinical Psychology 7: 755-765 (2012)
Evolution of cognitive functions | 9 months
  The evolution of cognitive functions will be assess with the Cambridge Neuropsychological Test Automated Battery (CANTAB).
  The CANTAB cognitive tests will be assess prior to intervention and then at month 3 and month 9 after the beginning of the intervention.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Epileptology Department of The Grenoble University Hospital, Grenoble
  - Epileptology Department of the Lyon University Hospital, Lyon
  - La Teppe medical centre, Tain-l'Hermitage

IPD SHARING:
Plan to Share IPD: No